CLINICAL TRIAL: NCT06181370
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, PK and PD of Inhaled AGMB-447 in Healthy Participants and Participants With Idiopathic Pulmonary Fibrosis
Brief Title: Phase I Study to Assess Safety, Tolerability, PK and PD of AGMB-447 in Healthy Participants and Participants With IPF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Agomab Spain S.L. (Industry)
Responsible Party: Sponsor
Organization: Agomab Therapeutics NV (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGMB-447-C101
Record Dates: First submitted 2023-12-11; First posted 2023-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: IPF

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGMB-447 (Experimental): Participants will receive a single dose of AGMB-447 (part A), multiple doses of AGMB-447 over 7 days (part B) or multiple doses of AGMB-447 over 14 days (part C)
  Interventions: Drug: AGMB-447
- placebo (Placebo Comparator): Participants will receive a single dose of placebo (part A), multiple doses of placebo over 7 days (part B) or multiple doses of placebo over 14 days (part C)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: AGMB-447 — AGMB-447 inhaled drug
  Arms: AGMB-447
Other: placebo — placebo inhaled drug
  Arms: placebo

SUMMARY:
The purpose of this study is to measure the safety, tolerability PK and PD of inhaled AGMB-477 compared with placebo in healthy participants and participants with IPF. This is an integrated phase 1, single center, 3-part, double-blind, randomized, placebo-controlled SAD (Part A) and MAD (Part B) study in healthy participants and multiple dose study in IPF participants (Part C).

Safety, tolerability PK and PD will be assessed following single ascending, multiple ascending and multiple dosing of AGMB-447 administered via nebulizer in Part A, B and C, respectively.

ELIGIBILITY:
Inclusion criteria for Healthy Participants (Parts A and B):

* Male and female participants aged between 18-55 years inclusive, at the time of informed consent.
* Participants must have FEV1 ≥80% predicted at screening and prior to randomization on Day -1 or Day 1 of treatment period 1 (using Global Lung Index, GLI 2012, predicted values).
* Participant must have a body weight of at least 50.0 kg and BMI ≥ 18 and ≤ 32 kg/m2 at screening.
* Participants must be in good health as determined by medical history, physical examination, vital signs, 12-lead ECG, spirometry and clinical laboratory assessments at the time of screening, as judged by the Investigator.

Inclusion Criteria for IPF Participants (Part C)

* Male and female participants aged >40 years inclusive, at the time of informed consent.
* Participants must have a confirmed diagnosis of IPF (IPF based on 2022 ATS/ERS/JRS/ALAT Guidelines) as confirmed by the Investigator based on chest High Resolution Computed Tomography Scan taken within 5 years of screening and, only if available, surgical lung biopsy)
* Participants must be either:
* Receiving a stable, well tolerated dose of Nintedanib for 3 months prior to screening for the treatment of IPF
* OR
* Receiving no current antifibrotic medication for the treatment of IPF. This includes those who have never received treatment and those who have stopped medication due to intolerance for any reason, except non-responsiveness, for at least 6 weeks prior to screening.
* Participants must have FVC ≥40% of predicted (using Global Lung Index, GLI 2012, predicted values) at screening.
* Participants must have DLCO (corrected for hemoglobin ) ≥ 25% of predicted (using Global Lung Index, GLI 2017, predicted values) at screening.
* Participants must have FEV1 ≥30% predicted at screening and prior to randomization on Day -1 or Day 1 (using Global Lung Index, GLI 2012, predicted values).

Exclusion criteria for Healthy Participants (Parts A and B)

* History or presence of any clinically relevant acute or chronic medical or psychiatric condition that could interfere with the participant's safety during the clinical study or expose the participant to undue risk as judged by the Investigator.
* After a minimum of 10 minutes supine rest at the time of screening or prior to randomization on Day -1 or Day 1 of treatment period 1:

  * Systolic blood pressure <90 or >150 mmHg, or
  * Diastolic blood pressure <50 or >95 mmHg, or
  * Pulse <40 or >90 bpm
* Any clinically significant abnormalities in resting ECG at the time of screening or prior to randomization on Day -1 or Day 1 of treatment period 1 including prolonged QTcF (>450 ms for males; >470 ms for females using the mean of triplicate ECG's) and cardiac arrhythmias, as judged by the Investigator.
* Clinically significant abnormalities in renal function at screening including any of the following:

  * Serum creatinine >2 x ULN
  * eGFR <80 mL/min
* Clinically significant abnormalities in liver function at screening including any of the following:

  * Bilirubin >1.5 x ULN
  * Aminotransferases >2 x ULN
  * ALP >1.5 x ULN

Exclusion Criteria for IPF Participants (Part C)

* History or presence of any clinically relevant acute or chronic medical or psychiatric condition that could interfere with the participant's safety during the clinical study or expose the participant to undue risk as judged by the Investigator.
* History or presence of any clinically significant pulmonary abnormalities, with the exception of IPF, in the opinion of the Investigator.
* Relevant airways obstruction (pre-bronchodilator FEV1/ FVC < 0.7) at screening.
* Any clinically significant abnormalities in resting ECG at the time of screening or prior to randomization on Day -1 or Day 1 including prolonged QTcF (>450 ms for males; >470 ms for females using the mean of triplicate ECG's) and cardiac arrhythmias, as judged by the Investigator.
* Clinically significant abnormalities in liver function at screening including any of the following:

  * Bilirubin >1.5 x ULN
  * Aminotransferases >2 x ULN
  * ALP >1.5 x ULN
* Acute IPF exacerbation within 3 months prior to screening and/or during the screening period prior to dose on Day 1 as determined by the Investigator.
* Any signs of respiratory tract infection within 4 weeks of screening or prior to dosing on Day 1 that is deemed clinically significant in the opinion of the Investigator.
* Malignancy within the past 5 years of screening with the exception of in situ removal of basal cell carcinoma or resected benign colonic polyps.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | From Screening Through Study Completion, up to 8 Weeks
  To evaluate the safety and tolerability of AGMB-447 in terms of AE at every visit
Number of participants with abnormal clinical laboratory values | From Screening Through Study Completion, up to 8 Weeks
  To evaluate the safety and tolerability of AGMB-129 in terms of abnormal laboratory parameters at every visit
Number of participants with abnormal ECG parameters | From Screening Through Study Completion, up to 8 Weeks
  To evaluate the safety and tolerability of AGMB-447 in terms of abnormal ECGs at every visit
Number of participants with abnormal vital signs | From Screening Through Study Completion, up to 8 Weeks
  To evaluate the safety and tolerability of AGMB-447 in terms of vital signs at every visit
Number of participants with abnormal physical exams | From Screening Through Study Completion, up to 8 Weeks
  To evaluate the safety and tolerability of AGMB-447 in terms of physical exams at every visit
Number of participants with abnormal spirometry parameters | From Screening Through Study Completion, up to 8 Weeks
  To evaluate the safety and tolerability of AGMB-447 in terms of spirometry at every visit

SECONDARY OUTCOMES:
Plasma levels of AGMB-447 | From Screening Through Study Completion, up to 8 Weeks
  To characterize the pharmacokinetics (PK) of AGMB-447 by measuring the amount in plasma
Plasma levels of the major metabolite | From Screening Through Study Completion, up to 8 Weeks
  To characterize the pharmacokinetics (PK) of the major metabolite by measuring the amount in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Wiesel, MD, Study Director — Agomab Therapeutics
Locations (1):
- Medicines Evaluation Unit Ltd. an IQVIA business, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No